CLINICAL TRIAL: NCT01146015
Title: Immunogenicity, Reactogenicity and Safety of the Trivalent Influenza Subunit Vaccine Influvac® for the Season 2010/2011. An Open-Label, Baseline-Controlled Multi-Center Study in Two Groups: Adult Subjects and Elderly Subjects
Brief Title: Annual Study to Investigate Inactivated Subunit Influenza Vaccine Due to New Virus Strains for the 2010/2011 Season
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Biologicals (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Organization: Abbott (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S201.3.130; 2010-018350-13 (EudraCT Number)
Record Dates: First submitted 2010-06-14; First posted 2010-06-17 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Influenza
Keywords: Influenza; Vaccine; CHMP criteria
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Trivalent influenza subunit vaccine Influvac

INTERVENTIONS:
Biological: Trivalent influenza subunit vaccine Influvac — 3x 15mcg HA per 0.5 ml,trivalent one injection at Day 1

SUMMARY:
Influenza (flu) viruses change continuously, therefore also the parts of viruses used in influenza vaccines can vary from year to year. In Europe, manufacturers/marketing holders of these vaccines are required to be involved in ongoing clinical trials and to present the results to the competent authorities each year. The current study is a phase IIIa clinical trial with a commercially available vaccine (Influvac®) supplied in pre filled syringes. It is part of the ongoing clinical trial program for Influvac® and will be done to assess the immunogenicity and safety and tolerability of next season's trivalent influenza subunit vaccine in two groups of subjects in good health: subjects aged >= 18 and <= 60 years and subjects >= 61 years of age (elderly)

ELIGIBILITY:
Inclusion Criteria

1. Willing and able to give informed consent and able to adhere to all protocol required study procedures.
2. Men and women aged >= 18 and <= 60 years or >= 61 years of age at the day of study vaccination.
3. Being in good health as judged by medical history, physical examination and clinical judgment of the investigator

Exclusion Criteria

1. Known to be allergic to eggs, chicken protein, gentamicin or any other constituent of the vaccine.
2. A serious adverse reaction after a previous (influenza) vaccination.
3. Presence of any significant condition that may prohibit inclusion as determined by the investigator.
4. Seasonal or pandemic influenza vaccination or laboratory confirmed seasonal or pandemic influenza infection within the previous six months before study vaccination or planned vaccination during the study period.
5. A history of Guillain-Barré syndrome or active neurological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2010-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
HI titers and its derived parameters after 2 weeks (seroprotection, seroconversion and mean fold increase), reactogenicity and inconvenience of Influvac® 2010/2011 as defined by the CHMP guideline for influenza vaccines | 2 weeks
HI titers and its derived parameters after 3 weeks (seroprotection, seroconversion and mean fold increase), reactogenicity and inconvenience of Influvac® 2010/2011 as defined by the CHMP guideline for influenza vaccines | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hanka de Voogd, MD, Study Director — Abbott Healthcare Products B.V.
Locations (2):
- Site Reference ID/Investigator# 44974, Tessenderlo, Belgium
- Site Reference ID/Investigator# 44975, Hamburg, Germany